CLINICAL TRIAL: NCT06840145
Title: Biomarkers of Neurodegeneration and Neuroplasticity in Parkinson's Disease Patients Treated by Intermittent Theta-burst Stimulation Over the Bilateral Primary Motor Area: A Randomized, Double-blind, Sham-controlled, Crossover Trial Study
Brief Title: Biomarkers of Neurodegeneration and Neuroplasticity in Parkinson's Disease Patients Treated by Bilateral M1-iTBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de investigación e innovación biomédica de Cádiz (Other)
Collaborators: Ministry of Science and Innovation, Spain (Other Government); Andalusian Ministry of Health and Families (Unknown); Andalusian Ministry of University, Research and Innovation (Unknown); University of Cadiz (Other); Hospital Universitario Puerta del Mar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PD-iTBS-2169-N-19
Record Dates: First submitted 2023-09-02; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Each patient received both active and sham iTBS in randomized order in two different sessions, separated by at least 3 months. All patients will be tested four times: at baseline (pre-stimulation) and after iTBS (post-stimulation), both for active and sham iTBS. In each session, motor evaluation will be performed at different follow-up visits along with a comprehensive neurocognitive assessment, evaluation of M1 excitability, combined structural MRI and resting-state EEG and fMRI, and serum biomarker quantification of neuroaxonal damage, astrocytic reactivity, and neural plasticity prior to and after iTBS.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The patient and the examiner who administered the clinical scales and all assessments were blind to the type of iTBS delivered, which was applied by another blinded experimenter.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- real iTBS (Active Comparator): Intermittent theta burst stimulation (iTBS) will be performed using a 3 pulse bursts at 50 Hz repeated every 200 ms and delivered as short trains of 10 bursts lasting 2 s and an intertrain silence period of 8 s, for a total of 600 pulses (20 cycles of trains) and a total duration of 190 s. Intensity of iTBS will be administered to the bilateral M1 at 80% of the active motor threshold (aMT) of each patient.
  Interventions: Device: repetitive transcranial magnetic stimulation
- sham iTBS (Sham Comparator): The repetitive transcranial magnetic stimulation (rTMS) coil stimulation will be applied in the same position of the real stimulation. Sham stimulation during treatment will follow the same procedure and both coils are identical in appearance and produce a similar sound and sensation, although the sham coil delivers no stimulation. The patient will hear the same sound of real stimulation, which will be only functionally inactive but will be completely performed (for the whole time of duration of stimulation)
  Interventions: Device: repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation — Intermittent theta Burst stimulation will be performed as detailed in the Real arm description
  Other Names: rTMS; intermittent theta-burst stimulation; iTBS

SUMMARY:
Intermittent theta-burst stimulation (iTBS) is a promising therapeutic option for Parkinson's disease patients. A study involving 24 patients will assess its effectiveness in alleviating clinical deficits. Patients will undergo 5 sessions of iTBS over the bilateral M1 and a 3-month washout period. Motor evaluation, neurocognitive assessment, serum biomarkers of neurodegeneration and neuroplasticity, and structural and functional MRI evaluations will be conducted at follow-up visits.

DETAILED DESCRIPTION:
Background and objectives:

Intermittent theta-burst stimulation (iTBS) is a patterned form of excitatory transcranial magnetic stimulation that has yielded encouraging results as an adjunctive therapeutic option to alleviate the emergence of clinical deficits in Parkinson's disease (PD) patients. Although it has been demonstrated that iTBS influences dopamine-dependent cortico-striatal plasticity, little research has examined the neurobiological mechanisms underlying iTBS-induce clinical enhancement. Here, the primary goal is to verify whether iTBS bilaterally delivered over the primary motor cortex (M1) is effective at reducing both scoring motor functioning and non-motor symptoms in PD. The investigators hypothesize that these clinical improvements following bilateral M1-iTBS could be driven by endogenous dopamine release, which may rebalance cortical excitability and restore compensatory striatal volume changes, resulting in increased striatal-cortical-cerebellar functional connectivity, and positively impacting neuroglia and neuroplasticity modification.

Methods:

A total of 24 PD patients will be assessed in a crossover, randomized, double-blind, sham-controlled protocol study involving application of iTBS over the bilateral M1 (M1 iTBS). Patients on medication will be randomly assigned to receive real iTBS or control (sham) stimulation and will undergo 5 sessions (1 week) of iTBS over the bilateral M1 (1 week), a 3-month washout period, and then 5 sessions (1 week) of sham stimulation. Motor evaluation will be performed at different follow-up visits along with a comprehensive neurocognitive assessment, evaluation of M1 excitability, combined structural magnetic resonance imaging (MRI) and resting-state electroencephalography and functional MRI, and serum biomarker quantification of neuroaxonal damage, astrocytic reactivity, and neural plasticity prior to and after iTBS.

Discussion:

The findings of this study will help to update the efficiency of M1 iTBS for the treatment of PD and further provide specific neurobiological insights into improvements in motor and nonmotor symptoms in these patients. This novel project aims to yield more detailed structural and functional brain evaluations using a noninvasive approach, with the potential to identify prognostic neuroprotective biomarkers and elucidate structural and functional mechanisms of M1 iTBS-induced plasticity in cortico-basal ganglia circuitry. The current approach may significantly optimize neuromodulation paradigms to ensure state-of-the-art and scalable rehabilitative treatment to alleviate motor and nonmotor symptoms of PD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with PD according to the UK Parkinson's Disease Society Brain Bank diagnostic criteria (UK PDSBB) diagnostic criteria
* Disease duration of at least 5 years to reduce the risk of including levodopa-responsive atypical Parkinsonism patients;
* Disease symptomatology in the ON medication state at a H&Y scale of II-III;
* Clinical and therapeutic stability in the last 2 months previous to the recruitment period; and
* Aged 45-75 years.

Exclusion Criteria:

* Lack of a PD diagnosis that meets the UK PDSBB diagnostic criteria
* Presence of a serious systemic disease
* Presence of severe or moderate cognitive impairment comparable to dementia, as revealed by an MMP score of ≤ 24
* Any incapacitating psychiatric or other clinical condition that might affect the correct performance of this protocol, such as any dystonia and/or dyskinesia
* Patients who received amantadine within the previous 60 days
* Any sign of atypical parkinsonism, neurological comorbidities, or history of cranioencephalic traumatism or epilepsy or any other contraindication for receiving neurostimulation with TMS (e.g., intracranial magnetic implant, cardiac pacemaker)

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-02-12 (Actual); Study Completion 2024-04-12 (Actual)

PRIMARY OUTCOMES:
Clinical motor improvement | Changes from baseline to immediately after stimulation, after 1 week, after 2 weeks, and after 4 weeks.
  Movement Disorders Society (MDS) Unified Parkinson's Disease Rating Scale (UPDRS) Part III (MDS-UPDRS III). Part III assessed the motor signs of PD and was administered by the rater (Range 0-132). Part III contained 33 scores based on 18 items. For each question a numeric score was assigned between 0-4, where 0 = Normal, 1 = Slight, 2 = Mild, 3 = Moderate, 4 = Severe.
Changes on quality of life and motor complications | Changes from baseline to after stimulation.
  MDS-UPDRS (parts II - IV). Part II assessed motor experiences of daily living (Range 0-52). Part IV assessed motor complications and contained 6 items. Score range: 0-24, 4 and below is mild, 13 and above is severe

SECONDARY OUTCOMES:
Change in levodopa equivalent daily dose (LEDD) | Changes from baseline to after stimulation
  Change in Levodopa and Dopamine Equivalent Daily Dosages (LEDD). The dosages of these medications are calculated using standardized conversion factors to obtain LEDD. This outcome aims to measure any changes in the daily dosages of these medications over the course of the study or intervention.
Change in the Parkinson's Fatigue Scale (PFS-16) | Changes from baseline to after stimulation
  The PFS-16 is a 16-item patient-rated scale based on recent feelings and experiences over the past two weeks. Nine items address the impact of fatigue on daily functioning and activities, including socialization and work but not exercise specifically and seven items tap the presence or absence of the subjective experience of fatigue with an emphasis on the physical effects of fatigue. The scoring possibilities are 1 for "strongly disagree" and 5 for "strongly agree". Based on the total of the scores, an ordinal PFS score ranging from 16 to 80 will be applied.
Change in quality of life measured with the Parkinson Disease Questionnaire-39 (PDQ-39) | Changes from baseline to after stimulation
  Mobility impact as assessed by PDQ-39 mobility dimension (questions #1-10 from the total PDQ-39 questionnaire). Scores are on a 0-4 Likert Scale (lower scores equaling better quality of life), summed, and then transformed into the total PDQ-39 that ranges from 0-100. Lower scores represent better quality of life.
Screening of cognitive function by MMP | Changes from baseline to 2 weeks after stimulation
  Mini Mental Parkinson (MMP) is a brief questionnaire derived from the Mini Mental State Examination and used for the assessment of general cognitive function in PD patients. This test is evaluated on a maximum of 32 points. The presence of severe or moderate cognitive impairment comparable to dementia is indicated by a score of ≤ 24.
Screening of frontal lobe function related activities by Frontal Assessment Battery (FAB) | Changes from baseline to after stimulation
  Frontal Assessment Battery (FAB) is a short battery consisting of 6 subtests related to different frontal lobe functions. The maximum score to be obtained in this test is 18 points. To consider that the subject presents alterations in the frontal lobe and, therefore, altered executive functions, his score must be equal to or less than 11 points.
Screening of visuospatial memory by Benton Visual Retention Test (BVRT) | Changes from baseline to after stimulation
  Benton Visual Retention Test (BVRT) is a test used for the evaluation of visuospatial memory. In our protocol, we plan to use the multiple choice format of administration, which consists of stimulus presentation followed by concealment for immediate recognition of one item out of four answer options (specifically, the M form). The performance is scored 0-10 based on correct drawing reconstruction.
Beck Depression Inventory-II (BDI-II) | Changes from baseline to 2 weeks after stimulation
  In the BDI-II, a score of 0-13 indicates absence of depression, 14-19 mild depression, 20-28 moderate depression, and 29-63 severe depression.
Hamilton Rating Scale for Anxiety (HAM-A) | Changes from baseline to 2 weeks after stimulation
  In the HAM-A has a score range of 0 to 56, where higher scores are associated with higher severity anxiety.
Starkstein Apathy Scale (SAS) | Changes from baseline to 2 weeks after stimulation
  The SAS has 14 items, rated on a 4-point scale with higher values indicating more apathy
Scale for the Evaluation of Neuropsychiatric Disorders in Parkinson's Disease (SEND-PD) | Changes from baseline to 2 weeks after stimulation
  The SEND-PD is a 12-item scale divided into three subscales: psychotic symptoms, mood/apathy, and impulse control behaviors. Items are rated from 0 (not present) to 4 (very severe)
Parkinson's Psychosis Questionnaire (PPQ) | Changes from baseline to 2 weeks after stimulation
  The PPQ is a screening tool used to measure the frequency and severity of early signs and psychotic symptoms of PD and consists of six items, each rated from 1 (no symptoms) to 4 (extreme symptoms); the total score ranges from 6 to 24 points.
Frontal Systems Behavior Scale (FrSBe) | Changes from baseline to 2 weeks after stimulation
  The FrSBe is a self-report scale designed to assess the changes in behavior that may occur in relation to frontal system dysfunction. Each item is rated on a 1-5 Likert scale. Raw scores for the three subscales (Apathy, Disinhibition, and Executive Dysfunction) and the Total are reported as T scores.
Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease (QUIP) | Changes from baseline to 2 weeks after stimulation
  The QUIP is a screening questionnaire developed for the assessment of Impulsive-Compulsive Disorders (ICDs) and related behaviors. It uses a 5-point Likert scale (score 0-4 for each question) to gauge the frequency of behaviors. Scores for each ICDs and related disorder range from 0 to 16 and the total QUIP score for all ICDs and related disorders combined ranges from 0 to 112, with a higher score indicating greater severity (ie, frequency) of symptoms.
Center for Neurologic Study-Lability Scale (CNS-LS) | Changes from baseline to 2 weeks after stimulation
  The CNS-LS is a screening instrument composed of seven items that are scored by the patient according to the perceived frequency of pseudobulbar affect (PBA) episodes during the last week. A CNS-LS score of 13 or higher may suggest PBA.
Cortical excitability TMS-EMG measures | Changes from baseline to immediately after stimulation
  The following transcranial magnetic stimulation (TMS)-derived measures of cortical excitability using electromyography (EMG) parameters of cortical excitability will be obtained after stimulation of the first dorsal interosseous (FDI) muscle hotspot of the mapping grid: the resting motor threshold (rMT); the active motor threshold (aMT); twenty single pulses ("20t"); and the cortical silent period (cSP)

OTHER OUTCOMES:
Resting-state EEG activity | Changes from baseline to 3 days after stimulation
  Power spectral density (PSD) analysis of delta, theta, alpha, beta, gamma rhythms, and functional connectivity measures (e.g., coherence, synchronization measures from graph theory metrics) of EEG signal recorded during eyes-closed (4 min) and eyes-open (4 min) conditions
Structural MRI - T1-weighted (T13D) | Changes from baseline to 1 week after stimulation
  Measures of global and regional gray matter (GM) volume and cortical thickness (CT) changes in magnetic resonance imaging (MRI) by voxel-based morphometry (VBM) measures
Resting-state functional fMRI | Changes from baseline to 1 week after stimulation
  Using baseline iTBS resting-state functional magnetic resonance imaging (fMRI), altered brain networks associated with PD will be identified by independent component analysis (ICA) and Seed-to-voxel and seed-to-seed functional connectivity measures between patients and controls.
Serum protein quantification of Neurofilament light (NfL) protein | Changes from baseline to 1 week after stimulation
  Quantification of serum NfL levels by Single-molecule assay (Simoa; SR-X™ biomarker detection system)
Serum protein quantification of Glial Fibrillary Acid Protein (GFAP) | Changes from baseline to 2 weeks after stimulation
  Quantification of serum GFAP levels by Single-molecule assay (Simoa; SR-X™ biomarker detection system)
Serum protein quantification of Brain-Derived Neurotrophic Factor (BDNF) | Changes from baseline to 2 weeks after stimulation
  Quantification of serum BDNF levels by Single-molecule assay (Simoa; SR-X™ biomarker detection system)

CONTACTS AND LOCATIONS:
Overall Officials: Javier J. Gonzalez-Rosa, PhD, Principal Investigator — University of Cadiz & Institute of Biomedical Research Cadiz (INiBICA)
Locations (1):
- Hospital Universitario Puerta del Mar, Cadiz, Cadiz, Spain

IPD SHARING:
Plan to Share IPD: Yes
The anonymized raw data analyzed in the present study are available on reasonable request to the corresponding author for purposes of replicating procedures and results.
  The Results derived from the project will be published in clinical and neuroscience journals.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Once the main results of the study have been published
Access Criteria: The anonymized raw data analyzed in the present study are available on reasonable request.

REFERENCES:
- [Derived] Rashid-Lopez R, Macias-Garcia P, Cruz-Gomez AJ, Cano-Cano F, Sanchez-Fernandez FL, Sarrias-Arrabal E, Del Marco A, Gonzalez-Moraleda A, Lozano-Soto E, Sanmartino F, Espinosa-Rosso R, Gonzalez-Rosa JJ. Plasticity-Induced Motor Recovery of Bilateral Intermittent Theta Burst Stimulation in Parkinson's Disease: A Randomized, Double-Blind, Sham-Controlled, Crossover Trial. Neurol Ther. 2026 Feb;15(1):345-366. doi: 10.1007/s40120-025-00865-0. Epub 2025 Dec 6. PMID 41351806